CLINICAL TRIAL: NCT00955422
Title: Screening and Evaluation of Patients With Signs and Symptoms of Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090198; 09-M-0198
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-07-06

CONDITIONS: Alzheimer's Disease
Keywords: Diagnosis; Alzheimer's Disease; Memory Disorder; Dementia; Alzheimer Disease; Memory Loss
MeSH Terms: conditions — Alzheimer Disease; Disease; Memory Disorders; Dementia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Individuals who demonstrate symptoms of Alzheimer s disease, such as progressive memory loss, may be eligible to participate in National Institutes of Health research studies. However, other physical and psychological conditions may produce symptoms similar to those of Alzheimer s disease. To determine whether a patient meets the eligibility criteria to participate in a research protocol, researchers must perform a series of diagnostic tests and procedures.
* These evaluations are designed to evaluate a participant s general medical condition (for example, blood tests and neurological exams) and to confirm a diagnosis or rule out an individual for consideration. They maximize the safety for participants in studies conducted at the National Institutes of Mental Health.

Objective:

- To determine the eligibility of individuals for active Alzheimer s disease protocols.

Eligibility:

- Individuals 45 years of age and older who have been having memory problems that have been getting worse with time and have been interfering with everyday life.

Design:

* Required tests and procedures for various research studies may include the following:
* Medical history and physical examination, including a psychiatric evaluation.
* Neuropsychological tests to test memory, mood, concentration, and thought processes.
* Blood and urine tests.
* Imaging studies (X-rays, magnetic resonance imaging (MRI), computerized tomography (CT), positron emission tomography (PET)).
* Additional blood samples and MRI data for future use.
* After all eligibility assessments are complete, participants may be offered participation in one or more research protocols

DETAILED DESCRIPTION:
Objective: To provide a mechanism for recruitment and screening of AD patients for inclusion into studies conducted at the National Institutes of Health. To provide data from MRI and [18F]FDG and PIB PET imaging from healthy volunteers to compare to that from AD patients. To provide longitudinal data from MRI and [18F]FDG and PIB PET imaging from both AD patients and healthy volunteers.

Study population: Patients with signs and symptoms of Alzheimer s disease. Healthy age-matched volunteers.

Design: Patients with signs and symptoms of Alzheimer s disease will be recruited from the community using advertisements and through communication with neurologists, psychiatrists, and general practitioners in the community. Patients will come to the NIH for an evaluation that may include medical and neurological evaluation, laboratory testing, brain MRI, neuropsychological evaluation, and brain imaging with [18F]fluorodeoxyglucose ([18F]FDG) and carbon-11 labeled Pittsburgh Compound B (PIB) PET. The focus of this protocol will be on assisting with the diagnosis of AD vs. another cause of memory impairment. Eligible patients will be offered participation in other protocols with the Molecular Imaging Branch. Eligible patients may also be referred to other studies at the NIH. Patients will not be offered treatment or long-term follow-up in this protocol. Age matched healthy volunteers will undergo brain imaging with MRI and with [18F]FDG and PIB PET. Healthy volunteers and patients who meet diagnostic criteria for AD will be asked to repeat study procedures after an interval of at least one year but no more than 5 years.

Outcome measures: Results from medical and neurological evaluation, neuropsychological testing, laboratory tests, and brain MRI will be used to determine if patients meet NINDS criteria for probable Alzheimer s disease. In patients who undergo brain imaging with [18F]FDG and PIB PET, PET data will be used for investigational purposes in subjects who participate in other protocols with the Molecular Imaging Branch. Results from brain imaging from healthy volunteers will be used to compare to that from AD patients. [18F]FDG and PIB PET may also be useful for determining if patients meet criteria for probable Alzheimer s disease.

ELIGIBILITY:
* Patients with signs and symptoms of Alzheimer s disease will be recruited from neurological and psychiatric clinics, from self or family referral in response to advertisements or from private physicians. Healthy volunteers will be recruited by the MIB.

INCLUSION CRITERIA:

1. Patients and healthy volunteers must be age 45 or older.
2. Patients must have a history of progressive memory impairment.
3. Patients must have a caregiver who is willing to accompany the subject to the NIH.

EXCLUSION CRITERIA FOR PATIENTS:

1. The diagnosis of a different type of dementia, including frontotemporal dementia, normal pressure hydrocephalus, Lewy body dementia, Parkinson s disease dementia, Huntington s disease, or vascular dementia.
2. Pregnant women. Women of childbearing potential will be screened by history for the possibility of pregnancy and undergo a urine pregnancy test.
3. Any medical contraindication to the procedures performed in the study, or any current severe medical or psychiatric illness other than Alzheimer s disease.
4. Behavioral symptoms that would preclude the gathering of data for the study, or advanced disease such that subjects cannot provide assent.

EXCLUSION CRITERIA FOR CONTROLS:

1. The diagnosis of a brain disorder.
2. Pregnant women.
3. Any medical contraindication to the procedures performed in the study, or any current severe medical or psychiatric illness.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2009-07-31; Study Completion 2017-07-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gorshow S. Alzheimer's disease and managed care: a convincing case for action. Manag Care Interface. 2007 Mar;20(3):26-7. PMID 17458478
- [Background] Wimo A, Jonsson L, Winblad B. An estimate of the worldwide prevalence and direct costs of dementia in 2003. Dement Geriatr Cogn Disord. 2006;21(3):175-81. doi: 10.1159/000090733. Epub 2006 Jan 9. PMID 16401889
- [Background] Dubois B, Feldman HH, Jacova C, Dekosky ST, Barberger-Gateau P, Cummings J, Delacourte A, Galasko D, Gauthier S, Jicha G, Meguro K, O'brien J, Pasquier F, Robert P, Rossor M, Salloway S, Stern Y, Visser PJ, Scheltens P. Research criteria for the diagnosis of Alzheimer's disease: revising the NINCDS-ADRDA criteria. Lancet Neurol. 2007 Aug;6(8):734-46. doi: 10.1016/S1474-4422(07)70178-3. PMID 17616482
- [Derived] Kreisl WC, Lyoo CH, Liow JS, Snow J, Page E, Jenko KJ, Morse CL, Zoghbi SS, Pike VW, Turner RS, Innis RB. Distinct patterns of increased translocator protein in posterior cortical atrophy and amnestic Alzheimer's disease. Neurobiol Aging. 2017 Mar;51:132-140. doi: 10.1016/j.neurobiolaging.2016.12.006. Epub 2016 Dec 16. PMID 28068564
- [Derived] Kreisl WC, Lyoo CH, Liow JS, Wei M, Snow J, Page E, Jenko KJ, Morse CL, Zoghbi SS, Pike VW, Turner RS, Innis RB. (11)C-PBR28 binding to translocator protein increases with progression of Alzheimer's disease. Neurobiol Aging. 2016 Aug;44:53-61. doi: 10.1016/j.neurobiolaging.2016.04.011. Epub 2016 Apr 27. PMID 27318133